CLINICAL TRIAL: NCT00076752
Title: A Pilot Study of Intensified Lymphodepletion Followed by Autologous Hematopoietic Stem Cell Transplantation in Patients With Severe Systemic Lupus Erythematosus
Brief Title: Lymphocyte Depletion and Stem Cell Transplantation to Treat Severe Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Pavletic, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040095; 04-C-0095; NCT00726518 (obsolete NCT alias)
Record Dates: First submitted 2004-02-02; First posted 2004-02-03 (Estimated); Results first posted 2014-06-10 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Refractory SLE; Immunoablation; Immunological Recovery; Efficacy; Mechanism of Disease; Lupus; Systemic Lupus Erythematosus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — fludarabine phosphate; Cyclophosphamide; Rituximab; Filgrastim; Methylprednisolone; Immunologic Techniques; Diphenhydramine; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous HSCT in SLE (Experimental): Autologous hematopoietic stem cell transplantation (HSCT) in systemic lupus erythematosus (SLE).
  SLE is a chronic, inflammatory disease of the immune system. Participants received a priming, conditioning and transplant regimen. Priming regimen consisted of treatment with rituxan, filgrastim, cyclophosphamide, mesna, fludarabine phosphate, and methylprednisolone. Conditioning and transplant regimen consisted of fludarabine, cyclophosphamide, rituxan, filgrastim, mesna, diphenhydramine and stem cell transplant infusion.
  Interventions: Drug: fludarabine phosphate; Drug: cyclophosphamide; Biological: Rituxan (rituximab); Biological: filgrastim; Drug: methylprednisolone; Other: immunologic technique; Other: laboratory biomarker analysis; Procedure: autologous hematopoietic stem cell transplantation; Drug: Diphenhydramine; Drug: Mesna

INTERVENTIONS:
Drug: fludarabine phosphate — Conditioning and transplant regimen: 30 mg/m^2 day intravenous infusion over 30 minutes daily, 4 days (transplant days -6, -5, -4, -3)
  Other Names: Fludara
Drug: cyclophosphamide — Priming regimen: 2000 mg/m^2 intravenous infusion over 2 hours, day 2. Conditioning and transplant regimen: 1200 mg/m^2 day intravenous infusion daily, 4 days (-6, -5, -4, -3).
  Other Names: Cytoxan
Biological: Rituxan (rituximab) — Priming regimen: 375 mg/m^2 intravenous day 1, 4. Conditioning and transplant regimen: 750 mg/m^2 intravenous infusion, day -7.
  Other Names: Rituximab
Biological: filgrastim — Priming regimen: 10 micrograms/kg/day subcutaneous, starting day 6. Conditioning and transplant regimen: 5 micrograms/kg/day subcutaneous, day +1 until ANC >500 microliters.
  Other Names: GCSF (growth colony stimulating factor)
Drug: methylprednisolone — Priming regimen:1000 mg intravenous over 30 minutes, day 1.
  Other Names: Medrol
Other: immunologic technique — Lymphoablative regimen using cyclophosphamide, rituximab, and fludarabine followed by a CD34 cell selected autologous stem cell transplant.
Other: laboratory biomarker analysis — Standard human immunology research laboratory ex vivo studies.
Procedure: autologous hematopoietic stem cell transplantation — Day 0, product will be infused rapidly intravenously after premedication with diphenhydramine 25-60 mg orally or intravenous.
Drug: Diphenhydramine — Conditioning and transplant regimen 25-50 mg orally or intravenously.
  Other Names: Benadryl
Drug: Mesna — Priming regimen: 600 mg/m^2 intravenous immediately prior to cyclophosphamide and repeat at 4 and 7 hours after the first dose, day 2. Conditioning and transplant regimen:1200 mg/m^2 per day continuous 24 hour intravenous infusion, daily for 4 days, start concurrently with the start of cyclophosphamide.
  Other Names: Mesnex

SUMMARY:
This study will examine a new approach to treating patients with severe systemic lupus erythematosus (SLE) that involves collecting stem cells (cells produced by the bone marrow that develop into blood cells) from the patient, completely shutting down the patient's immune system, and then giving back the patient's stem cells. SLE is a chronic, inflammatory disorder of the immune system that can affect many organs. It is called an autoimmune disease because the patient's lymphocytes (white blood cells that normally protect against invading organisms), go out of control and attack the body's own tissues.

Patients between 15 and 40 years of age with severe SLE affecting a major organ that is resistant to standard treatment may be eligible for this study. Candidates are screened with a medical history and physical examination, blood and urine tests, skin tuberculin test, and radiology studies to evaluate the extent of disease. They have endocrinology, nutrition, dental, and social work consultations, ultrasound or MUGA (multi-gated acquisition scan) scan heart imaging, electrocardiogram and lung function tests, bone marrow biopsy, and lymph node aspirate. Depending on which organs are affected, patients may have additional tests, such as lumbar puncture (spinal tap), kidney or lung biopsy, MRI (magnetic resonance imaging) of the brain and spinal cord, and PET (positron emission tomography) scan. They also complete quality of life questionnaires and have disability functional testing and neurocognitive (thinking) assessments.

Participants have a central venous line (plastic tube) inserted into a neck or chest vein for administering stem cells and medicines and for drawing blood. They undergo seven apheresis procedures during the course of the study to collect stem cells for transplant and for research. For apheresis, whole blood is collected through a needle in an arm vein and directed to a cell-separating machine where the white cells are extracted and the rest of the blood is returned to the patient through the same needle.

Patients are primed with three medications (methylprednisolone, rituximab, and cyclophosphamide) through the central line to help control the disease. In addition, a medication called G-CSF (growth colony stimulating factor) is injected under the skin for several days to boost production of stem cells. After enough stem cells have been collected for transplantation (infusion through the central line), patients are admitted to the hospital for an 8-day conditioning regimen followed by transplantation. The conditioning treatment consists of rituximab, fludarabine, and cyclophosphamide to eliminate all the white blood cells from the blood and bone marrow. The stem cells are then infused and the patient is closely monitored by a team of physicians and nurses. When the stem cells have engrafted, the bone marrow has recovered, and the patient feels well enough - usually 2 to 3 weeks after transplant - the patient is discharged from the hospital. Prednisone tapering begins as soon as feasibly possible, but no later then 28 days after transplant.

Patients return to the National Institutes of Health (NIH) Clinical Center for frequent follow-up visits during the first 2 to 3 months following transplant. The time between visits is then extended to once every 3 months the first year, then every 6 months the second year, and then at least yearly for 5 years after the transplant. These visits include a physical examination, blood and urine tests, lumbar puncture (if there is central nervous system involvement), other appropriate biopsies and tests as needed to monitor the patient's health, short apheresis procedures to collect blood for research purposes, and quality of life questionnaires. Some select procedures will be optional. Bone marrow biopsies and lymph node aspirates are done at beginning and at 6, 12, and 24 months after transplant. PET scans are done at 1, 6, 12, and 24 months.

...

DETAILED DESCRIPTION:
Background:

* Systemic lupus erythematosus (SLE) is a systemic autoimmune disease that can involve almost any organ and can range in severity from mild to life-threatening. In spite of significant improvements in survival of SLE patients over last 20 years, a small but significant portion of patients still develop progressive therapy-refractory disease that impairs organ function and overall survival.
* Since 1996, more than 500 patients have been treated worldwide in pilot trials of autologous hematopoietic stem cell transplantation (autoHSCT) for autoimmune diseases, including about 80 patients with SLE.
* The rationale for autoHSCT in autoimmune disease is to ablate autoreactive immune effectors and allow reconstitution of a new self-tolerant immune system from the

hematopoietic stem cell. Studies have demonstrated acceptable safety and promising short term efficacy of high-dose cyclophosphamide-based (200 mg/kg) autoHSCT for about 60% of patients with advanced refractory SLE and reacquisition of sensitivity to conventional drugs have been demonstrated in many cases. However, these trials were designed to address the primary endpoint of safety and were inadequate for assessing the disease response.

-Numerous questions about the true efficacy of autoHSCT, optimal transplant regimen, patient selection and mechanisms of action remain unaddressed.

Objectives:

* The primary objective is to assess the rate of continuous relapse-free complete clinical responses at 24 months post-transplant, with statistical power of 84% to detect, if greater than 70 percent of patients meet the primary endpoint.
* The long-term goal of this research is to develop a basis for future transplant protocols that would incorporate new cellular or other immunotherapeutic interventions to further improve results of transplants with the ultimate goal to cure SLE.

Eligibility:

-Subjects age 15-40 years who fulfill at least 4 of the 11 criteria for SLE as defined by the

American College of Rheumatology

-Have severe and active lupus, refractory to immunosuppressive therapy. Included are subjects with nephritis, central nervous system (CNS) lupus, pulmonary lupus or hematologic disease

Design:

* Fourteen patients with active and standard dose cyclophosphamide-resistant SLE will be enrolled on this phase II pilot study.
* Study design is intended to improve the efficacy of autoHSCT. A lymphoablative conditioning regimen (rituximab, fludarabine and cyclophosphamide) is explored for the first time in autoimmune disease.
* The treatment schedule consists of two parts; the priming regimen prior to stem cell mobilization and collection, and the conditioning regimen with transplant.
* In contrast to other studies, this study has precisely defined eligibility and disease response criteria with strict schema of tapering immunosuppression that should allow accurate interpretation of the treatment results.
* The study includes a carefully chosen battery of laboratory research studies designed to investigate SLE biology and mechanisms of post-transplant responses.

ELIGIBILITY:
-INCLUSION CRITERIA

1. Age 15-40 years
2. Must fulfill at least 4 of the following 11 criteria for systemic lupus erythematous (SLE) as defined by the American College of Rheumatology:

   -Malar rash. Fixed erythema, flat or raised, over the malar eminences, tending to spare the nasolabial folds.
   * Discoid rash. Erythematous raised patches with adherent keratotic scaling and follicular plugging; atrophic scarring may occur in older lesions.
   * Photosensitivity. Skin rash as a result of unusual reaction to sunlight, by patient history or physician observation.
   * Oral ulcers. Oral or nasopharyngeal ulcerations, usually painless, observed by a physician.
   * Arthritis. Nonerosive arthritis involving two or more peripheral joints, characterized by tenderness, swelling, or effusion.
   * Serositis. a.) Pleuritis - convincing history of pleuritic pain or rub heard by a physician or evidence of pleural effusion

   OR

   b.) Pericarditis - documented by electrocardiogram (ECG) or rub or evidence of pericardial effusion

   -Renal disorder. a.) Persistent proteinuria greater than 0.5 grams per day or greater than 3+ if quantitation not performed

   OR

   b.) Cellular casts - may be red cell, hemoglobin, granular, tubular, or mixed.
   * Neurologic disorder. a.) Seizures - in the absence of offending drugs or known metabolic derangements; eg, uremia, ketoacidosis, or electrolyte imbalance

   OR

   b.) Psychosis - in the absence of offending drugs or known metabolic derangements; eg, uremia, ketoacidosis, or electrolyte imbalance

   -Hematologic disorder. a.) Hemolytic anemia - with reticulocytosis

   OR

   b.) Leukopenia - less than 4000/ L total on two or more occasions

   OR

   c.) Lymphopenia - less than 1500/ L on two or more occasions

   OR

   d.) Thrombocytopenia - less than 100,000/ L in the absence of offending drugs
   * Immunologic disorder. a.) Anti-deoxyribonucleic acid (DNA): antibody to native DNA in abnormal titer

   OR

   b.) Anti-SM: presence of antibody to SM nuclear antigen

   OR

   c.) Positive finding of antiphospholipid antibodies based on (1) an abnormal serum level of immunoglobulin G (IgG) or immunoglobulin M (IgM) anti-cardiolipin antibodies, (2) a positive test result for lupus anticoagulant using a standard method, or (3) false positive serologic test for syphilis known to be positive for at least 6 months and confirmed by Treponema Pallidum immobilization or fluorescent treponemal antibody absorption test

   -Antinuclear antibodies. An abnormal titer of ANAs by immunofluorescence or an equivalent assay at any point in time in the absence of drugs known to be associated with drug-induced lupus syndrome.
3. Have severe and active lupus, refractory to immunosuppressive therapy, defined as one of the following (a-d):

   a.Nephritis: Biopsy proven Diffuse Proliferative Glomerulonephritis (World Health Organization (WHO) Class IV) with or without superimposed membranous changes

   i.Active disease:

<!-- -->

1. A kidney biopsy within three months of enrollment showing active WHO Class IV disease. Activity will be determined based on the presence of endocapillary cellular proliferation compromising the capillary loops or cellular crescents or necrosis on light microscopy or subendothelial deposits on electron microscopy.
2. If a biopsy is contraindicated patients can be enrolled if they had a previous biopsy showing Diffuse Proliferative Glomerulonephritis (WHO Class IV) and at the time of enrollment have all of the following:

   1. Proteinuria greater than 1gm/day
   2. Active urine sediment defined as hematuria (greater than 10 red blood cell (RBC)/hpf (high power field) on a nephrology urinalysis of a 50 mL urine sample) with dysmorphic RBC and/or cellular casts on a nephrology urinalysis of a 50 mL urine sample
   3. Low C3 (less than 69 mg/dL) and/or elevated dsDNA antibodies (greater than 25EU)
3. Need for prednisone greater than 20 mg/day due to increased renal activity after at least 6 months of cyclophosphamide.

ii. Treatment resistant:

1. Patients with active disease after at least 6 months of intravenous pulse cyclophosphamide +/- iv methylprednisolone and daily oral prednisone, or
2. Early flare: those who have reactivation of their nephritis during or within 6 months of completing cyclophosphamide therapy
3. Recalcitrant disease: two or more recurrences of lupus nephritis within five years of enrollment. All flares must have received adequate therapy and least one of the episodes must have been treated with minimum 6 months of intravenous pulse cyclophosphamide plus iv methylprednisolone and maintenance oral prednisone.

   Central nervous system (CNS) lupus: Lupus CNS manifestations indicative of encephalitis or myelitis or vasculitis. Concomitant CNS diseases should be excluded. (e.g. infections, multiple sclerosis; patients fulfilling multiple sclerosis (MS) and SLE criteria will be excluded). Clinical signs and symptoms must be supported by objective findings of CNS inflammation.

   i. Active disease:

   Signs/symptoms that are accepted for disease activity:

   -Clinical signs and symptoms compatible with focal CNS damage -Severe global neurocognitive/psychiatric impairment (eg: psychosis, organic brain syndrome, severe depression)

   -Intractable seizures

   Clinical findings must be supported by at least one of the following:
   1. Magnetic resonance imaging (MRI) findings consistent with transverse myelitis or

      Central nervous system (CNS) vasculitis

      - Signs of inflammation on MRI are either the presence of Gadolinium (Gd)-enhancing lesions, or the increase of the number and/or volume of T2-weighted lesions (or lesions showing up on fluid attenuated inversion recovery (FLAIR) imaging). We will use the standard MS protocol sequences, which are routinely used in the Clinical Center to evaluate inflammatory CNS lesions.
   2. If patient has seizures/psychiatric signs and symptoms in the absence of clear signs of vasculitis or cerebritis by MRI, the cerebral spinal fluid (CSF) should show protein elevation above normal levels and abnormal number of white blood cells (WBCs) or intrathecal IgG synthesis/or oligoclonal bands.
   3. Need for prednisone greater than 20 mg/day due to increased CNS activity (see above) after at least three months of cyclophosphamide therapy.

   ii-Treatment resistant:

   a) Active disease after a minimum of three months of oral or intravenous cyclophosphamide, or

   b) Early flare: reactivation of CNS lupus within 6 months of completing cyclophosphamide therapy

   c. Recalcitrant disease: two or more recurrences of CNS lupus within five years of enrollment. All flares must have received adequate therapy and at least one of the episodes must have been treated with minimum three months of oral or intravenous cyclophosphamide.

   Pulmonary lupus

   i. Active disease:
   1. Lung biopsy showing active pneumonitis, alveolitis or pulmonary vasculitis after the minimally required therapy within one month of enrollment or
   2. If a biopsy is contraindicated within one month of enrollment, patients may be included if they had a biopsy at the start or during cyclophosphamide treatment showing active pneumonitis, alveolitis or pulmonary vasculitis (as above) and have abnormal or worsening pulmonary function tests with a chest computed tomography (CT) consistent with active pneumonitis, alveolitis or vasculitis within 2 weeks of enrollment and at the time of enrollment have a CT consistent with active disease.
   3. Need for prednisone greater than 20 mg/day due to increased pulmonary lupus activity after minimum of three months of cyclophosphamide.

      ii. Treatment resistant:
   4. Ongoing or recurrent active pulmonary lupus after a minimum of three months of oral or intravenous cyclophosphamide, or
   5. Early flare: reactivation of pulmonary lupus (as defined above) within 6 months of completing cyclophosphamide therapy.
   6. Recalcitrant disease: two or more recurrences of pulmonary as described above within five years of enrollment. All flares must have received adequate therapy and at least one of the episodes must have been treated with minimum 3 months of oral or intravenous cyclophosphamide.

   i) Active disease:

   a) Severe immune-mediated thrombocytopenia (platelet count less than 20,000/mm^3 or less than 50,000/mm^3 with history of bleeding), or

   b) Severe immune-mediated anemia (requiring transfusions to maintain hemoglobin (Hb) greater than 8.0 g/dL or to treat symptoms of anemia) c) Need for prednisone greater than 20 mg/day due to increased hematologic lupus activity after therapy as described in section ii.a).

   ii) Treatment resistant:

   a) Active disease as defined above after a minimum of three months of high dose oral or pulse corticosteroids +/- intravenous immunoglobulin (IVIg) (or WinRho) and splenectomy, or

   b) Early flare: reactivation of hematologic lupus (as defined above) within 6 months of completing above therapy.

   c) Recalcitrant disease: two or more recurrences of immune-mediated thrombocytopenia or anemia, as described above, within five years of enrollment. All flares must have received adequate therapy and at least one of the episodes must have been treated by splenectomy.

   EXCLUSION CRITERIA

1. Inability to provide written informed consent prior to entry in the protocol

2. Pregnant or lactating women. Women of childbearing potential are required to have a negative pregnancy test at screening

3. Women of childbearing potential who are not practicing or who are unwilling to practice birth control during the entire study

4. Men who are unwilling to practice birth control for the first 6 months after the transplant

5. Evidence of infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)

6. History of malignancy other than basal cell carcinoma of the skin

7. Carbon monoxide diffusing capacity (DLCO) corrected less than 45%

8. Left ventricular ejection fraction (LVEF) less than 45%, determined by ECHO cardiogram or MUGA

9. Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) greater than 2x upper limit of normal (unless active myopathy is proven by elevation of serum aldolase levels and the patient has no obvious hepatic disease) and/or bilirubin greater than 2.0 (unless due to isolated hemolysis).

10. Calculated glomerular filtration rate less than 30 ml/min using the modification of diet in renal disease (MDRD) equation estimate:

Glomerular filtration rate (GFR) (ml/min/173 m^2) =186.3 x (Pcr) exponential -1.154 x (age) exponential -0.203 x 1.212 (if black) x 0.742 (if female)

11. Late flare (patients who have target organ flare, that is not within the time frame defined as early flare, will not be considered as treatment failures until they receive the minimally required therapy for this flare episode and fail to respond to it)

12. Abnormal bone marrow cytogenetics

13. Significant concurrent medical condition or any significant circumstance that could affect the patient's ability to tolerate or complete the study

14. Live vaccines within 4 weeks of starting the priming regimen

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2004-01-30; Primary Completion 2013-10-15 (Actual); Study Completion 2013-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Pavletic, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shlomchik MJ, Craft JE, Mamula MJ. From T to B and back again: positive feedback in systemic autoimmune disease. Nat Rev Immunol. 2001 Nov;1(2):147-53. doi: 10.1038/35100573. PMID 11905822
- [Background] Manzi S, Meilahn EN, Rairie JE, Conte CG, Medsger TA Jr, Jansen-McWilliams L, D'Agostino RB, Kuller LH. Age-specific incidence rates of myocardial infarction and angina in women with systemic lupus erythematosus: comparison with the Framingham Study. Am J Epidemiol. 1997 Mar 1;145(5):408-15. doi: 10.1093/oxfordjournals.aje.a009122. PMID 9048514
- [Background] Lipsky PE. Systemic lupus erythematosus: an autoimmune disease of B cell hyperactivity. Nat Immunol. 2001 Sep;2(9):764-6. doi: 10.1038/ni0901-764. No abstract available. PMID 11526379
- [Result] Illei GG, Cervera R, Burt RK, Doria A, Hiepe F, Jayne D, Pavletic S, Martin T, Marmont A, Saccardi R, Voskuyl AE, Farge D. Current state and future directions of autologous hematopoietic stem cell transplantation in systemic lupus erythematosus. Ann Rheum Dis. 2011 Dec;70(12):2071-4. doi: 10.1136/ard.2010.148049. Epub 2011 Aug 26. PMID 21873334
- [Derived] Goklemez S, Hasni S, Hakim FT, Muraro PA, Pirsl F, Rose J, Memon S, Fowler DF, Steinberg SM, Baker EH, Panch SR, Gress R, Illei GG, Lipsky PE, Pavletic SZ. Long-term follow-up after lymphodepleting autologous haematopoietic cell transplantation for treatment-resistant systemic lupus erythematosus. Rheumatology (Oxford). 2022 Aug 3;61(8):3317-3328. doi: 10.1093/rheumatology/keab877. PMID 34875023

RESULTS

PARTICIPANT FLOW:
Groups:
- Autologous HSCT in SLE: Autologous hematopoietic stem cell transplantation (HSCT) in systemic lupus erythematosus (SLE).
  SLE is a chronic, inflammatory disease of the immune system. Participants received a priming, conditioning and transplant regimen. Priming regimen consisted of treatment with rituxan, filgrastim, cyclophosphamide, mesna, fludarabine phosphate, and methylprednisolone. Conditioning and transplant regimen consisted of fludarabine, cyclophosphamide, rituxan, filgrastim, mesna, and diphenhydramine. Stem cell transplant infusion day 0, product will be infused rapidly intravenously after premedication with diphenhydramine 25-60 mg orally or intravenous.
Period: Overall Study
Arm/Group | Autologous HSCT in SLE
Started | 9
Completed | 6
Not Completed | 3
Not completed — Death | 2
Not completed — Withdrawal per PI, PI put study on hold | 1

BASELINE CHARACTERISTICS:
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.85 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Relapse-free Complete Clinical Response
Description: Complete clinical response is defined as complete clinical response in the target organ and no clinical signs of active lupus as determined by a Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) score of ≤3; prednisone ≤10mg/day at 6 months and ≤5mg/day at 12 months or later.
Time Frame: 60 months
Population: Ninth participant was taken off study before proceeding with transplant per principal investigator due to decision to put study on hold.
Measure: Median (Full Range); unit: Months
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 8
Months | 54 [36 to 60]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 9
participants | 8

3. Secondary Outcome: Anti-Nuclear Antibody
Description: Anti-Nuclear antibody is a well accepted biological clinical laboratory marker of systemic lupus. Range of normal values is 0-0.9 EU.
Time Frame: Day -7, day 0, 1 3, and 6 months, 1 year, 18 months, 2 years and 3 years.
Population: One participant was enrolled but the study was closed before the patient could be treated.
Measure: Mean (Standard Deviation); unit: EU
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 8
EU
  Day -7 | 5.4 (4.65)
  Day 0 | 4.7 (4.73)
  1 month | 3.7 (3.89)
  3 months | 3.2 (3.91)
  6 months: number analyzed (Participants) | 7
  6 months | 2.7 (3.01)
  1 year: number analyzed (Participants) | 5
  1 year | 2.6 (2.77)
  18 months: number analyzed (Participants) | 5
  18 months | 2.8 (2.7)
  2 years: number analyzed (Participants) | 5
  2 years | 2.5 (2.59)
  3 years 9: number analyzed (Participants) | 4
  3 years 9 | 2.5 (2.96)

4. Secondary Outcome: Extractable Nuclear Antigen (ENA)
Description: Extractable nuclear antigen is a well accepted biological clinical laboratory marker of systemic lupus. Range of normal values is 0-19.
Time Frame: Day -7, day 0, 1 3, and 6 months, 1 year, 18 months, 2 years and 3 years.
Population: One participant was enrolled but the study was closed before the patient could be treated.
Measure: Mean (Standard Deviation); unit: EU
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 8
EU
  Day -7 | 66.9 (74.48)
  Day 0 | 64.8 (70.61)
  1 month | 61.5 (73.72)
  3 months | 58.5 (67.03)
  6 months: number analyzed (Participants) | 7
  6 months | 51.3 (57.22)
  1 year: number analyzed (Participants) | 5
  1 year | 57.2 (58.07)
  18 months: number analyzed (Participants) | 5
  18 months | 60.6 (60.76)
  2 years: number analyzed (Participants) | 5
  2 years | 50.6 (49.04)
  3 years: number analyzed (Participants) | 3
  3 years | 26.3 (41.12)

5. Secondary Outcome: Anti-Double Stranded Deoxyribonucleic Acid (DNA) Antibody
Description: Anti-Double stranded deoxyribonucleic acid antibody is a well accepted biological clinical laboratory marker especially specific for systemic lupus. Range of normal values is 0-24 IU.
Time Frame: Day -7, day 0, 1 3, and 6 months, 1 year, 18 months, 2 years and 3 years.
Population: One participant was enrolled but the study was closed before the patient could be treated.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 8
IU
  Day -7 | 17.3 (24.92)
  Day 0 | 8.8 (16.8)
  1 month | 0 (0)
  3 months | 0 (0)
  6 months: number analyzed (Participants) | 7
  6 months | 0 (0)
  1 year: number analyzed (Participants) | 5
  1 year | 0 (0)
  18 months: number analyzed (Participants) | 5
  18 months | 0 (0)
  2 years: number analyzed (Participants) | 5
  2 years | 0 (0)
  3 years: number analyzed (Participants) | 5
  3 years | 0 (0)

6. Secondary Outcome: Anti-Smith-Ribonuclear Protein Antibody
Description: Anti-Smith-Ribonuclear protein antibody is a well accepted biological clinical laboratory marker of systemic lupus.Range of normal values is 0-19 EU.
Time Frame: Day -7, day 0, 1 3, and 6 months, 1 year, 18 months and 2 years.
Population: One participant was enrolled but the study was closed before the patient could be treated.
Measure: Mean (Standard Deviation); unit: EU
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 5
EU
  Day -7 | 49 (49.51)
  Day 0 | 51.6 (53.72)
  1 month: number analyzed (Participants) | 4
  1 month | 31.5 (40.31)
  3 months | 29.8 (41.48)
  6 months: number analyzed (Participants) | 4
  6 months | 28.5 (40.07)
  1 year: number analyzed (Participants) | 3
  1 year | 20 (34.64)
  18 months: number analyzed (Participants) | 3
  18 months | 16.67 (28.87)
  2 years: number analyzed (Participants) | 3
  2 years | 25.67 (44.46)

7. Secondary Outcome: White Blood Cells
Description: The white blood cell test was performed to investigate immunological efficacy and mechanisms of response after lymphodepleting auto-hematopoietic stem cell transplant for systemic lupus erythematosus. Range of normal values is 3.4-9.6 K/uL.
Time Frame: Day -7, day 0, 1 3, and 6 months, 1 year, 18 months, 2 years and 3 years.
Population: One participant was enrolled but the study was closed before the patient could be treated.
Measure: Mean (Standard Deviation); unit: K/uL
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 8
K/uL
  Day -7 | 6.89 (3.07)
  Day 0 | 0.47 (0.31)
  1 month | 10.32 (6.6)
  3 months | 3.84 (1.4)
  6 months: number analyzed (Participants) | 7
  6 months | 4.21 (1.38)
  1 year: number analyzed (Participants) | 5
  1 year | 5.81 (1.01)
  18 months: number analyzed (Participants) | 5
  18 months | 5.24 (0.82)
  2 years: number analyzed (Participants) | 5
  2 years | 7.17 (3.93)
  3 years: number analyzed (Participants) | 5
  3 years | 6.34 (1.08)

8. Secondary Outcome: Absolute Neutrophil Count
Description: The absolute neutrophil count test was performed to investigate immunological efficacy and mechanisms of response after lymphodepleting auto-hematopoietic stem cell transplant for systemic lupus erythematosus. Range of normal values is 1.29-7.5 K/uL.
Time Frame: Day -7, day 0, 1 3, and 6 months, 1 year, 18 months, 2 years and 3 years.
Population: One participant was enrolled but the study was closed before the patient could be treated.
Measure: Mean (Standard Deviation); unit: K/uL
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 8
K/uL
  Day -7 | 5.66 (2.88)
  Day 0 | 0.45 (0.3)
  1 month | 9.11 (6.67)
  3 months | 2.72 (0.93)
  6 months: number analyzed (Participants) | 7
  6 months | 2.78 (1.38)
  1 year: number analyzed (Participants) | 5
  1 year | 3.44 (0.97)
  18 months: number analyzed (Participants) | 5
  18 months | 2.72 (1.04)
  2 years: number analyzed (Participants) | 5
  2 years | 4.04 (1.7)
  3 years: number analyzed (Participants) | 5
  3 years | 3.77 (0.63)

9. Secondary Outcome: Absolute Lymphocyte Count
Description: The absolute lymphocyte count test was performed to investigate immunological efficacy and mechanisms of response after lymphodepleting auto-hematopoietic stem cell transplant for systemic lupus erythematosus. Range of normal values is 0.45-4.9 K/uL.
Time Frame: Day -7, day 0, 1 3, and 6 months, 1 year, 18 months, 2 years and 3 years.
Population: One participant was enrolled but the study was closed before the patient could be treated.
Measure: Mean (Standard Deviation); unit: K/uL
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 8
K/uL
  Day -7 | 0.54 (0.4)
  Day 0 | 0.0065 (0.0064)
  1 month | 0.42 (0.18)
  3 months | 0.53 (0.46)
  6 months: number analyzed (Participants) | 7
  6 months | 0.82 (0.31)
  1 year: number analyzed (Participants) | 5
  1 year | 1.75 (0.64)
  18 months: number analyzed (Participants) | 5
  18 months | 1.8 (0.61)
  2 years: number analyzed (Participants) | 5
  2 years | 1.8 (0.84)
  3 years: number analyzed (Participants) | 5
  3 years | 1.75 (0.56)

10. Secondary Outcome: Platelet Count
Description: The platelet count test was performed to investigate immunological efficacy and mechanisms of response after lymphodepleting auto-hematopoietic stem cell transplant for systemic lupus erythematosus. Range of normal values is 162-380 K/uL.
Time Frame: Day -7, day 0, 1 3, and 6 months, 1 year, 18 months, 2 years and 3 years.
Population: One participant was enrolled but the study was closed before the patient could be treated.
Measure: Mean (Standard Deviation); unit: K/uL
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 8
K/uL
  Day -7 | 251 (62.9)
  Day 0 | 113 (49)
  1 month | 166 (61.6)
  3 months | 187 (95.4)
  6 months: number analyzed (Participants) | 7
  6 months | 170 (64)
  1 year: number analyzed (Participants) | 5
  1 year | 226 (47.9)
  18 months: number analyzed (Participants) | 5
  18 months | 210 (43.5)
  2 years: number analyzed (Participants) | 5
  2 years | 308 (251.5)
  3 years: number analyzed (Participants) | 5
  3 years | 272 (125.4)

11. Secondary Outcome: Cluster of Differentiation 3 (CD3) + Cells
Description: The CD3+Cells test was performed to investigate immunological efficacy and mechanisms of response after lymphodepleting auto-hematopoietic stem cell transplant for systemic lupus erythematosus. Range of normal values is 650-2108 uL.
Time Frame: Day 0, 1 month, 3 months, 6 months, 1 year and 2 years.
Population: One participant was enrolled but the study was closed before the patient could be treated.
Measure: Mean (Standard Deviation); unit: cells/mL^3
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 8
cells/mL^3
  Day 0 | 2.99 (3.25)
  1 month | 239.47 (210.74)
  3 months | 435.97 (335.69)
  6 months: number analyzed (Participants) | 7
  6 months | 699.47 (256.67)
  1 year: number analyzed (Participants) | 6
  1 year | 1493.29 (605.26)
  2 years: number analyzed (Participants) | 5
  2 years | 1678.76 (888.41)

12. Secondary Outcome: Cluster of Differentiation 4 (CD4) + Cells
Description: The CD4 + Cells test was performed to investigate immunological efficacy and mechanisms of response after lymphodepleting auto-hematopoietic stem cell transplant for systemic lupus erythematosus. Range of normal values is 358-1259 uL.
Time Frame: Day 0, 1 month, 3 months, 6 months, 1 year and 2 years.
Population: One participant was enrolled but the study was closed before the patient could be treated.
Measure: Mean (Standard Deviation); unit: cells/mL^3
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 8
cells/mL^3
  Day 0 | 2.58 (2.98)
  1 month | 103.37 (117.43)
  3 months | 112.8 (101.94)
  6 months: number analyzed (Participants) | 7
  6 months | 316.25 (193.01)
  1 year: number analyzed (Participants) | 6
  1 year | 702.87 (362.75)
  2 years: number analyzed (Participants) | 5
  2 years | 958.03 (735.04)

13. Secondary Outcome: Cluster of Differentiation 8 (CD8) + Cells
Description: The CD8 + Cells test was performed to investigate immunological efficacy and mechanisms of response after lymphodepleting auto-hematopoietic stem cell transplant for systemic lupus erythematosus. Range of normal values is 194-836 u/L.
Time Frame: Day 0, 1 month, 3 months, 6 months, 1 year and 2 years.
Population: One participant was enrolled but the study was closed before the patient could be treated.
Measure: Mean (Standard Deviation); unit: cells/mL^3
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 8
cells/mL^3
  Day 0 | 0.34 (0.34)
  1 month | 138.68 (112.61)
  3 months | 318.47 (259.28)
  6 months: number analyzed (Participants) | 7
  6 months | 334.91 (139.55)
  1 year: number analyzed (Participants) | 6
  1 year | 736.67 (532.19)
  2 years: number analyzed (Participants) | 5
  2 years | 674.69 (378.6)

14. Secondary Outcome: Cluster of Differentiation 19 (CD19) + Cells
Description: The CD19 + Cells test was performed to investigate immunological efficacy and mechanisms of response after lymphodepleting auto-hematopoietic stem cell transplant for systemic lupus erythematosus. Range of normal values is 47-409 u/L.
Time Frame: Day 0, 1 month, 3 months, 6 months, 1 year and 2 years.
Population: One participant was enrolled but the study was closed before the patient could be treated.
Measure: Mean (Standard Deviation); unit: cells/mL^3
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 8
cells/mL^3
  Day 0 | 0.01 (0.02)
  1 month | 0.23 (0.32)
  3 months | 6.7 (17.22)
  6 months: number analyzed (Participants) | 7
  6 months | 45.32 (58.21)
  1 year: number analyzed (Participants) | 6
  1 year | 142.69 (116.24)
  3 years: number analyzed (Participants) | 5
  3 years | 246.83 (316.53)

15. Secondary Outcome: Natural Killer Cells
Description: The natural killer cells test was performed to investigate immunological efficacy and mechanisms of response after lymphodepleting auto-hematopoietic stem cell transplant for systemic lupus erythematosus. Range of normal values is 87-505 uL.
Time Frame: Day 0, 1 month, 3 months, 6 months, 1 year and 2 years.
Population: One participant was enrolled but the study was closed before the patient could be treated.
Measure: Mean (Standard Deviation); unit: cells/mL^3
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 8
cells/mL^3
  Day 0 | 0.03 (0.035)
  1 month | 117.06 (81.76)
  3 months | 116.57 (93.57)
  6 months: number analyzed (Participants) | 7
  6 months | 123.18 (63.32)
  1 year: number analyzed (Participants) | 6
  1 year | 158.9 (136.42)
  3 years: number analyzed (Participants) | 5
  3 years | 115.18 (68.3)

16. Secondary Outcome: Systemic Lupus Erythematosus Disease Activity Index (SLEDAI)
Description: The SLEDAI activity index test was performed to investigate immunological efficacy and mechanisms of response after lymphodepleting auto-hematopoietic stem cell transplant for systemic lupus erythematosus. Complete clinical response is defined as complete clinical response in the target organ and no clinical signs of active lupus as determined by a SLEDAI score of ≤3; partial response is at least 50% improvement in general disease activity as measured by SLEDAI. Remission is a SLEDAI score <3 and prednisone <10mg/day. 6+ indicates active disease requiring therapy. A score of 0 indicates a better outcome and a score greater then 6+ indicates a worse outcome.
Time Frame: Day -7, day 0, 1 month, 3 months, 6 months, 1 year, 18 months, 2 years and 3 years.
Population: One participant was enrolled but the study was closed before the patient could be treated.
Measure: Mean (Standard Deviation); unit: scores on a scale.
Arm/Group | Autologous HSCT in SLE
Number analyzed (Participants) | 8
scores on a scale.
  Day -7 | 4.25 (3.28)
  Day 0 | 4.13 (4.49)
  1 month | 3.63 (2.83)
  3 months: number analyzed (Participants) | 5
  3 months | 1.6 (3.58)
  6 months: number analyzed (Participants) | 4
  6 months | 0 (0)
  1 year: number analyzed (Participants) | 4
  1 year | 0 (0)
  18 months: number analyzed (Participants) | 2
  18 months | 0 (0)
  2 years: number analyzed (Participants) | 2
  2 years | 0 (0)
  3 years: number analyzed (Participants) | 2
  3 years | 0 (0)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Autologous HSCT in SLE
All-Cause Mortality (participants affected / at risk) | 2/9
Serious Adverse Events (participants affected / at risk) | 8/9
Other Adverse Events (participants affected / at risk) | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous HSCT in SLE (N=9)
allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
conduction abnormality/atrioventricular heart block: asystole (Cardiac disorders) | 1 (1)
hypertension (Cardiac disorders) | 1 (1)
gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 1 (1) — laparoscopic surgery w/appendectomy
infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with grades 3 or 4 neutrophils (ANC <1.0x10e9/L): lung (pneumonia)
infection - Other (Specify, CMV antigenemia without neutropenia) (Infections and infestations) | 1 (1)
ALT/SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1)
AST/SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1)
potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
encephalopathy (Nervous system disorders) | 1 (2)
hydrocephalus (Nervous system disorders) | 1 (2)
neuropathy: motor (Nervous system disorders) | 1 (1)
neuropathy: sensory (Nervous system disorders) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Death Not Associated with CTCAE term: Death NOS (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous HSCT in SLE (N=9)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1 (1)
Auditory/Ear - Other (Specify, __) (Ear and labyrinth disorders) | 1 (1) — hearing diminished on the left side
Blood/Bone Marrow - Other (Specify, __) (Blood and lymphatic system disorders) | 1 (2) — low HGB (anemia); low HGB
Bone marrow cellularity (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 8 (55)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 8 (82)
Lymphopenia (Blood and lymphatic system disorders) | 8 (79)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 8 (81)
Platelets (Blood and lymphatic system disorders) | 8 (130)
Supraventricular and nodal arrhythmia:: Atrial fibrillation (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia:: Supraventricular arrhythmia NOS (Cardiac disorders) | 1 (3)
Ventricular arrhythmia:: PVCs (Cardiac disorders) | 1 (1)
Ventricular arrhythmia:: Ventricular tachycardia (Cardiac disorders) | 1 (1)
Cardiac General - Other (Specify, __) (Cardiac disorders) | 1 (7) — 2+L leg edema; 2+ pitting R leg edema; 3+ pitting L leg edema; 3+ pitting edema R leg; intermittent 2+, 3+ pitting b/l LE edema
Cardiac troponin I (cTnI) (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 4 (4)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 4 (8)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) — (e.g., thrombotic thrombocytopenic purpura [TTP] or hemolytic uremic syndrome [HUS])
Constitutional Symptoms - Other (Specify,decreased appetite ) (General disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3 (8)
Rigors/chills (General disorders) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatology/Skin - Other (Specify, scalp dermatitis) (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (3)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 1 (1)
Masculinization of female (Endocrine disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (5)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (clinical exam):: Oral cavity (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (9)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (8)
Hemorrhage/Bleeding - Other (Specify,bruising-skin) (Blood and lymphatic system disorders) | 1 (1)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 2 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Febrile neutropenia (Infections and infestations) | 3 (4) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L):: Bladder (urinary)
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L):: Urinary tract NOS
Infection - Other (Specify, __) (Infections and infestations) | 2 (2) — R toe infection, was believed fungal; clostridium difficile in stool
Infection with normal ANC or Grade 1 or 2 neutrophils:: Abdomen NOS (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils:: Blood (Infections and infestations) | 4 (8)
Infection with normal ANC or Grade 1 or 2 neutrophils:: Bone (osteomyelitis) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils:: Catheter-related (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils:: Colon (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils:: Conjunctiva (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils:: Eye NOS (Infections and infestations) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils:: Lung (pneumonia) (Infections and infestations) | 2 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils:: Pharynx (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils:: Sinus (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils:: Small bowel NOS (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils:: Upper airway NOS (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils:: Urinary tract NOS (Infections and infestations) | 3 (4)
Infection with unknown ANC:: Middle ear (otitis media) (Infections and infestations) | 1 (1)
Infection with unknown ANC:: Urinary tract NOS (Infections and infestations) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 5 (36)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 5 (41)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5 (31)
Alkaline phosphatase (Metabolism and nutrition disorders) | 4 (25)
Amylase (Metabolism and nutrition disorders) | 3 (6)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 3 (8)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (6)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 8 (67)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 3 (9)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 5 (24)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (5)
Hemoglobinuria (Metabolism and nutrition disorders) | 3 (16)
Lipase (Metabolism and nutrition disorders) | 2 (5)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 3 (13)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 4 (10)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 7 (86)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 5 (16)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5 (14)
Proteinuria (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4 (8)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 2 (6)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (2)
Memory impairment (Nervous system disorders) | 1 (1)
Mood alteration:: Agitation (Nervous system disorders) | 1 (1)
Mood alteration:: Anxiety (Nervous system disorders) | 1 (1)
Mood alteration:: Depression (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 2 (2) — residual itching post herpetic area; episcleritis
Retinopathy (Eye disorders) | 1 (2)
Vision-blurred vision (Eye disorders) | 4 (4)
Vision-photophobia (Eye disorders) | 1 (1)
Pain - Other (Specify, __) (General disorders) | 1 (2) — b/l flanks; intermittent pain in hips and knees
Pain:: Abdomen NOS (Gastrointestinal disorders) | 2 (2)
Pain:: Back (Musculoskeletal and connective tissue disorders) | 5 (7)
Pain:: Bone (Musculoskeletal and connective tissue disorders) | 5 (7)
Pain:: Chest wall (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain:: Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain:: External ear (Ear and labyrinth disorders) | 1 (1)
Pain:: Eye (Eye disorders) | 2 (2)
Pain:: Head/headache (Nervous system disorders) | 5 (5)
Pain:: Muscle (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain:: Neck (Musculoskeletal and connective tissue disorders) | 3 (6)
Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 1 (2) — nasal congestion; nasal drainage
Cystitis (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-07-26): https://cdn.clinicaltrials.gov/large-docs/52/NCT00076752/Prot_SAP_000.pdf
  • Informed Consent Form (2006-01-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT00076752/ICF_001.pdf